CLINICAL TRIAL: NCT00248066
Title: APPRAISAL Trial: A Phase IIa Study to Evaluate the Safety and Preliminary Efficacy of RESTEN-MP® When Used in Conjunction With a Bare Metal Stent in de Novo Native Coronary Artery Lesions
Brief Title: Safety and Efficacy of RESTEN-MP When Used in Conjunction With a Bare Metal Stent in Coronary Arteries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Baim Institute for Clinical Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4126-17
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2007-02-08 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: Coronary artery disease; Restenosis; Coronary stent restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

INTERVENTIONS:
Drug: RESTEN-MP

SUMMARY:
The process of re-narrowing of a coronary artery following a revascularization procedure such as angioplasty, begins at the time of the procedure. Restenosis has long been considered a major problem for effective long-term interventional success. This often results in repeated procedures to deal with recurrent stenosis (or restenosis) of the original targeted vessel.

There is a substantial body of literature suggesting that local MYC protein production in the injured coronary artery is a major stimulus and potential cause of restenosis that appears after stent placement. This study is based upon the hypothesis that stopping MYC protein production in the vessel will help reduce restenosis (vessel re-narrowing).

AVI BioPharma Inc., has utilized its proprietary antisense chemistry to design a drug that interferes with MYC production.

This study will evaluate the safety and potential effectiveness of RESTEN-MP to reduce in-stent restenosis following balloon angioplasty and stent placement. The post-dose follow-up period is up to six-months.

RESTEN-MP is administered at the time a stent is successfully placed in a coronary artery, and again 24 hours later, via slow-push intravenous administration.

DETAILED DESCRIPTION:
The process of restenosis, the re-narrowing of a coronary artery lumen following a revascularization procedure, begins at the time of percutaneous coronary intervention (PCI). Restenosis has long been seen as a major impediment of effective long-term interventional cardiology, necessitating repeated procedures to deal with in situ recurrent stenosis of the original targeted vessel. The restenosis rates are between 30 to 50% of patients treated with balloon angioplasty and between 15 to 30% of patients treated with bare metal stents. There is currently high enthusiasm for drug-eluting stents already approved for the market and which have an overall restenosis rate of < 3% as reported in published reports for most clinical trial patient populations. However, there are subsets of patients (e.g., diabetic patients and patients with diffuse small vessel disease) that have restenosis rates around 10% despite the use of drug-eluting stents. It is probably too early to conclude that the currently approved drug-eluting stents are a panacea to relieve coronary arterial obstruction due to atherosclerotic heart disease. In fact, with the increased usage of the current drug-eluting stents on the market, there are reports of problems such as late stent malposition, subacute and late thromboses, and aneurysm formations due to the vessel toxicity associated with this method of treatment. There remains a definite need for a simple, safe and durable solution to restenosis.

The development of devices such as intravascular ultrasound has led to a greater understanding of restenosis mechanisms, especially after coronary artery stenting. It is presumed that the pathogenesis of coronary artery restenosis after a revascularization procedure entails two major processes. The first component (viz., recoil and remodeling) involves the mechanical collapse and constriction of the treated vessel; however, coronary stents provide luminal scaffolding that eliminates recoil and remodeling. The second component of coronary artery restenosis after a revascularization procedure is the endothelial response to injury. Whereas, the former focus in modulating the pathophysiological mechanisms involved in restenosis centered mainly on inhibition of platelet aggregation and function, current targets of pharmaceutical agents for this condition have shifted to inhibitors of the cell cycle, smooth muscle cell proliferation and migration, synthesis of extra-cellular matrix, and inflammatory mediators. Many different agents are currently being evaluated in pre-clinical and clinical studies.

AVI-4126, the active ingredient of RESTEN-MP, is a proprietary antisense drug designed to interrupt the translation of the human <c-myc> gene by mRNA. Therefore, the basis for this study is to ascertain if RESTEN-MP is safe and has a therapeutic benefit. Slow-push intravenous administration of RESTEN-MP in pharmacological doses in the restenosis porcine model prevented subsequent in-stent stenosis.

This clinical study will evaluate the safety and potential effectiveness of RESTEN-MP to reduce in-stent restenosis following balloon angioplasty. In order to objectively assess the therapeutic value of RESTEN-MP compared to other drugs used in combination with coronary artery stents and to utilize a sensitive method to assess the effectiveness of RESTEN-MP as a neointimal hyperplasia inhibitor, late loss between the time of stent placement and 6 months later is the therapeutic endpoint in this study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. An acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), coronary artery stenting, and emergent coronary artery bypass graft (CABG).
3. Clinical evidence of ischemic heart disease or a positive functional study.
4. The target lesion/vessel must meet the following criteria:

   1. The target lesion is a single de novo lesion that has not been previously treated with any interventional procedure. Only one lesion may be treated per subject.
   2. The target vessel must be a native coronary artery with a stenosis of ≥ 50% and < 100%.
   3. The target lesion must be ≥ 10 mm and ≤ 30 mm in length.
   4. The target vessel reference diameter must be ≥ 2.5 mm and ≤ 4.0 mm.
5. Female subjects of childbearing potential must have a documented negative serum pregnancy test within seven days before the procedure.
6. The subject or the subject's legally authorized representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.
7. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
8. The subject is capable of providing informed consent and has provided written consent prior to study entry.

Exclusion Criteria:

1. Documented left ventricular ejection fraction < 30%.
2. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, stainless steel, or sensitivity to contrast media, which cannot be adequately pre-medicated.
3. Evidence of an acute myocardial infarction within 72 hours of the intended treatment [defined as: Q wave or non-Q wave infarction having creatine kinase (CK) enzymes ≥ 2 times the upper laboratory normal (with the presence of a CK-MB elevated above the Institution's upper limit of normal)] or acute myocardial infarction in progress at time of treatment.
4. Previous coronary interventional procedure of any kind within the 30 days prior to the stent-placement procedure.
5. Planned interventional treatment of either the target or any non-target vessel within 30 days post-stent placement procedure is required.
6. Target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, or rotational atherectomy).
7. Previous stenting anywhere in the target vessel.
8. Target vessel has evidence of thrombus or is excessively tortuous (2 bends > 90° to reach the target lesion).
9. Target lesion has any one of the following characteristics:

   1. Lesion location is aorto-ostial, an unprotected left main lesion, or within 5 mm of the origin of the left anterior descending coronary artery (LAD), left circumflex coronary artery (LCX), or right coronary artery (RCA);
   2. Involves a side branch > 2.0 mm in diameter;
   3. Is at or distal to a 45º bend in the vessel; or
   4. Is moderately to severely calcified.
10. History of a stroke or transient ischemic attack within the prior 6 months.
11. Active peptic ulcer or has had upper gastrointestinal (GI) bleeding within the prior 6 months.
12. History of a bleeding diathesis or coagulopathy or will refuse blood transfusions.
13. Concurrent medical condition with a life expectancy of less than 12 months.
14. Any previous or planned treatment with other anti-restenosis therapies including, but not limited to, brachytherapy in the target vessel within 30 days of the stent placement procedure. [Note: Staged treatment of a non-target vessel is appropriate 30 days after enrollment.]
15. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. [Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.]
16. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-09

PRIMARY OUTCOMES:
Evaluate the potential efficacy of RESTEN-MP given intravenously upon confirmation of stent implantation and again at 24 hours post-stent implantation
The therapeutic endpoint to assess potential efficacy is the prevention of coronary late lumen loss 6 months after the stent placement procedure, based on quantitative coronary angiography (QCA).

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) defined as cardiac death, MI (Q wave and non-Q wave), emergent cardiac bypass surgery, and clinically-driven target lesion revascularization (TLR) at Days 14 and 30, and Month 6, 9 and 12 post-stent placement
Target vessel failure (TVF) rate, defined as a composite of target vessel revascularization, recurrent MI (Q or Non Q-Wave), or cardiac death that could not be clearly attributed to a vessel other than the target vessel at Month 9 post-stent placement
Angiographic binary restenosis (≥ 50% diameter stenosis) at Month 6 post-stent placement
In-stent minimum lumen diameter (MLD) at Month 6 post-stent placement
In-segment MLD at Month 6 post-stent placement
Proximal and distal late loss at Month 6 post-stent placement.
In-stent and in-segment percent (%) diameter stenosis at Month 6 post-stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sack, MD, Principal Investigator — Cardiac Clinic, University of Essen, Germany
Locations (3):
- Germany (3):
  - Coburg Hospital - Cardiology Clinic, Coburg
  - Cardiology Clinic, University Hospital of Essen, Essen
  - University Hospital of Heidelberg, Cardiology Clinic, Heidelberg